CLINICAL TRIAL: NCT05179668
Title: SGLT2 Inhibition (Dapagliflozin) in Diabetic and Non-diabetic Hemodialysis Patients With and Without Residual Urine Volume: a Prospective Randomized, Placebo-controlled, Double-blinded Phase II Trial
Brief Title: SGLT2 Inhibition in Hemodialysis
Acronym: DAPA-HD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Manfred Hecking, MD PhD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-Nr.: 1196/2021; 2021-000733-14 (EudraCT Number)
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Kidney Failure; Hemodialysis; Diabetes Mellitus, Type 2; Chronic Kidney Disease; Left Ventricular Hypertrophy
Keywords: Dapagliflozin; SGLT2 inhibition
MeSH Terms: conditions — Renal Insufficiency; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin 10 mg (Experimental)
  Interventions: Drug: Dapagliflozin 10 MG
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — administered orally once daily
  Other Names: Forxiga 10 MG
  Arms: Dapagliflozin 10 mg
Drug: Placebo — administered orally once daily
  Arms: Placebo tablet

SUMMARY:
Dapagliflozin will be compared with placebo to evaluate its effects on cardiac structure and safety in patients with kidney failure receiving maintenance hemodialysis.

DETAILED DESCRIPTION:
The Dapagliflozin in Hemodialysis (DAPA-HD) trial is an academic, multicenter, randomized, double-blind, placebo-controlled phase 2 study designed to assess the cardiovascular effects of dapagliflozin in patients with kidney failure undergoing maintenance hemodialysis. A total of 220 patients are randomized 1:1 to dapagliflozin 10 mg once daily or matching placebo for six months, with stratification according to residual urine output. The primary endpoint is the change in left ventricular mass indexed to body surface area, assessed by transthoracic echocardiography after six months of treatment. Secondary endpoints include additional echocardiographic measures, biomarker changes, quality of life, clinical events, and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Maintenance hemodialysis 3×/week for ≥ 3 months and ≤5 years
* BMI <45 kg/m2 and stable weight (±5 kg ["dry weight"]) over the preceding three months
* Interventricular septum width >11 mm

Exclusion Criteria:

* Treatment with SGLT2i within the last 6 months
* Hypersensitivity or Intolerance of SGLT2 inhibitors
* History of Type 1 diabetes mellitus
* History of diabetic ketoacidosis
* Scheduled kidney transplant from a living donor
* Acute coronary syndrome during the last 30 days
* Severe valvular heart disease
* Women of childbearing potential and unwilling or unable to use an acceptable method to avoid pregnancy for the entire study (estrogen and/or progesterone treatment).
* Pregnancy
* Breast feeding
* Substance abuse
* Life expectancy < 1 year
* Other significant disease or pathology, that might predispose that patient to an unacceptable risk or interferes with the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass indexed to body surface area | 6 months
  Change in left ventricular mass indexed to body surface area using echocardiography

SECONDARY OUTCOMES:
Change in left ventricular mass indexed to body height assessed by echocardiography | 6 months
Change in LVEF assessed by echocardiography | 6 months
Change in in LA volume index assessed by echocardiography | 6 months
Change in in GLS assessed by echocardiography | 6 months
Change in in Cardiac Biomarkers (NT-proBNP, hsTnT) | 6 months
Change in health-related quality of life | 6 months
Change in LV end-diastolic volume assessed by echocardiography | 6 months
Change in LV end-systolic volume assessed by echocardiography | 6 months
Change in body weight | 6 months
Change in blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hecking, MD, PhD, Principal Investigator — Medical University of Vienna, Department of Medicine III, Division of Nephrology and Dialysis; Thomas A Zelniker, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (9):
- Austria (9):
  - Dialyseinstitut Dr. Waller, Feldbach
  - Dialyseinstitut Gießauf GmbH, Graz
  - Klinik Landstraße, Vienna
  - Medical University of Vienna, Vienna
  - Klinik Favoriten, Vienna
  - Krankenhaus Hietzing, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinik Donaustadt, Vienna
  - Wiener Dialysezentrum, Vienna

IPD SHARING:
Plan to Share IPD: No